CLINICAL TRIAL: NCT06290154
Title: Factors Associated With Short-Term Major Adverse Cardiovascular Events After Liver Transplantation
Brief Title: Factors Associated With Posttransplant Cardiac Outcomes
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jia Liu, Dr, Sun Yat-sen University
Other Study IDs: RG2024-022-02
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Liver Transplantation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — clinical data and comprehensive echocardiography variables
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular disease has become the leading cause of death early after liver transplantation (LT). The aging LT population is accompanied with the increasing prevalence of cardiovascular risk factors such as hypertension, diabetes, and hyperlipidemia. Furthermore, cirrhosis has been known to cause alterations in the systemic haemodynamic system and cardiac muscle dysfunction, systolic and/or diastolic, known as Cirrhotic cardiomyopathy (CCM). Hence, transthoracic echocardiography is required in all LT candidates for preprocedural evaluation and risk stratification. However, traditional echocardiographic indices of cardiac function have low sensitivity. It is unclear whether comprehensive echocardiographic multiparameters, including speckle tracking echocardiograph (STE) and tissue doppler imaging (TDI) can help improve preoperative risk stratification. Therefore, we sought to analyze the ability of clinical and comprehensive echocardiography variables to predict intraoperative and perioperative cardiac events and cardiac mortality in our LT patient experience up to early post-liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* End-stage cirrhosis patients who will receive liver transplantation,
* Patients voluntarily take part in the study and write informed consent.

Exclusion Criteria:

* Decreased left ventricular systolic function (ejection fraction <45%),
* Significant uncorrectable structural cardiac abnormalities (eg, symptomatic coronary heart disease, advanced cardiomyopathy, severe valvular disease, severe congenital heart disease, etc),
* Uncontrolled pulmonary hypertension defined as pulmonary arterial systolic pressure ≧ 35mm Hg at rest despite maximal medical management,
* Circulatory or respiratory system with a score of 4 based on the preoperative Organ Dysfunction (CLIF-SOFA) score,
* Second-time liver transplantation,
* Combined organ transplantation,
* Satisfactory quality echocardiography could not be obtained before operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage cirrhosis who are going to undergo liver transplantation in the Third Affiliated Hospital of Sun Yat-sen University
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
a composite outcome of new cardiovascular disease after liver transplantation | 3 months after liver transplantation
  new symptomatic CAD, new heart failure (systolic and/or diastolic), new arrhythmia (atrial and/or ventricular), and/or new cardiac arrest, or cardiac death.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ren, Dr, Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (2):
- China (2):
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong